CLINICAL TRIAL: NCT05331287
Title: First Hospital of Qinhuangdao，Hebei Province, China
Brief Title: Comparing the "Snifing Position" , "Simple Head Extension" and "Neutral Position"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 5866
Record Dates: First submitted 2022-03-27; First posted 2022-04-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Therapeutic Procedural Complication
Keywords: Snifing Position; Simple Head Extension; neutral position; Nasotracheal intubation
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- snifing Position (Experimental): Nasotracheal intubation via fiberoptic bronchoscope under snifing position.The snifing position was obtained by placement of a 7-cm cushion under the head of the patient. When the FOB was inserted into Nasal cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB.
  Interventions: Other: Head position
- neutral position (Experimental): Nasotracheal intubation via fiberoptic bronchoscope under snifing position.The Head Extension was obtained by the occiput of the patient close to the operating table. When the FOB was inserted into Nasal cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB.
  Interventions: Other: Head position
- Head Extension (Experimental): Nasotracheal intubation via fiberoptic bronchoscope under snifing position.The extension position with a 7-cm pillow underneath the shoulder and the occiput close to the operating table. When the FOB was inserted into Nasal cavity, and the epiglottis and glottis were identified by the FOB. The anterior of FOB was inserted deep into tracheal after the glottis was exposed sufficiently then the tracheal tube was pushed into the trachea via the FOB.
  Interventions: Other: Head position

INTERVENTIONS:
Other: Head position — Influence of different head position on nasal endotracheal intubation

SUMMARY:
The simple head extension is recommended for optimization of glottic visualization during Nasotracheal intubation via fiberoptic bronchoscope (FOB) . However, no study confirmed its superiority over"snifing position" and "Neutral Position". In a prospective, randomized study, the authors compared the snifing position , simple head extension and "Neutral Position" in Nasotracheal intubation via fiberoptic bronchoscope.

DETAILED DESCRIPTION:
The study included ninety patients with anticipated difficult airways. The snifing position was obtained by placement of a 7-cm cushion under the head of the patient; the extension head position was obtained by placement of a 7-cm cushion under the shoulder; the neutral position with the occiput close to the operating table. The head position was randomized as follows: neutral position group (NP group), sniffing position group (SP group) or extension position group (EP group). Randomization (1:1:1) was based on the codes generated by Excel software, which were kept in sequentially numbered opaque envelopes until the began of study.

ELIGIBILITY:
Inclusion Criteria:

• ASA classifications of I-II, modified Mallampati classification of 3 or 4, requiring general anesthesia were included.

Exclusion Criteria:

* • ASA class IV or V

  * Abnormalities of the heart, brain, liver, lung, kidney and coagulation functions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Intubation Time | Ten minutes
  The primary endpoints were the time to view the vocal cords (TVC) which was taken when the operator indicated verbally that he view the vocal cords and the time to successful tracheal intubation (TSI). TSI was defined as the time taken from insertion of the FOB between the teeth until the appearance of a capnograhy curve.

SECONDARY OUTCOMES:
Occurrence of throat pain measured by VAS | one day Postoperative]

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Qinhuangdao, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: No